CLINICAL TRIAL: NCT02027402
Title: To Drain or Not to Drain in Laparoscopic Cholecystectomy for the Patients With Acutely Inflamed Gallbladder ; a Multicenter Randomized Controlled Trial
Brief Title: Effects of Drainage in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Assistant proffesor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: seoul -S2
Record Dates: First submitted 2013-12-30; First posted 2014-01-06 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Acute Cholecystitis; Empyema of Gallbladder; Abscess of Gallbladder
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drain insertion (Experimental): Laparoscopic cholecystectomy with drain insertion is performed in this arm.
  Interventions: Procedure: Laparoscopic cholecystectomy with drain insertion
- no drain insertion (No Intervention): In this arm, investigators perform only laparoscopic cholecystectomy, and not insert a drain

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy with drain insertion — In the drain insertion group, investigators use the closed suction drain through a lateral 5-mm trocar and placed it in right subhepatic space
  Arms: Drain insertion

SUMMARY:
During laparoscopic surgery for an acutely inflamed gallbladder, most surgeons routinely insert a drain. However, no consensus has been reached regarding the need for drainage in these cases, and the use of a drain remains controversial. This study is coordinated to find out the surgical outcomes and perioperative morbidity according to the insertion of drain after laparoscopic cholecystectomy. Investigators expect that the routine use of a drain after laparoscopic cholecystectomy for an acutely inflamed gallbladder will have no effects on the postoperative morbidity.

DETAILED DESCRIPTION:
Drain has been widely used in many abdominal surgeries for therapeutic purposes such as the removal of infected debris or abscess, and supporting the healing of leakage or fistula. Although the usability of therapeutic drain is commonly accepted, the efficacy of prophylactic drain still has been debated. Most surgeons have inserted prophylactic drain with expectations that the drain would be helpful for early detection of postoperative bleeding or leakage, and also prevention of intra-abdominal abscess through removing debris or curd. However, there are only few evidence-based studies for the actual effectiveness of prophylactic drain and the objections against the routine use of drain have been raised.

Most surgeons have placed the drain after cholecystectomy with expectations that it could help to detect postoperative bleeding or bile leakage and prevent intra-abdominal infection. However, there is a lack of evidence regarding the role of drain in laparoscopic cholecystectomy for acutely inflamed gallbladder and surgeons have placed the drain based on their experiences and beliefs, not on evidence-based guidelines. In the previous retrospective study, [4] we described that the routine drain use in laparoscopic cholecystectomy for acutely inflamed gallbladder has no advantage to detect bile leak or bleeding and it was no helpful to prevent the postoperative morbidities such as intra-abdominal abscess or wound infection. The aim of present multicenter trial is to assess the value of routine drain use in laparoscopic cholecystectomy for acutely inflamed gallbladder in a large, randomized controlled prospective study.

ELIGIBILITY:
Inclusion Criteria:

* acutely inflamed gallbladder

Exclusion Criteria:

* chronic cholecystitis
* gallbladder polyp or gallbladder cancer
* the patient who underwent reduced port surgery
* the patient who underwent common bile duct exploration during the operation
* the patient who underwent concurrent operation
* the patient who had past history of upper abdominal surgery
* the patient who had a immunodeficiency state
* the case which had a suspicion of delayed bile leakage
* the case which had a incomplete cystic duct ligation
* the patient who underwent open conversion surgery during the operation
* the patient who had a high risk of bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taeho Hong, Principal Investigator — SeoulSt.Mary's hospital
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

REFERENCES:
- [Derived] Kim EY, Lee SH, Lee JS, Yoon YC, Park SK, Choi HJ, Yoo DD, Hong TH. Is routine drain insertion after laparoscopic cholecystectomy for acute cholecystitis beneficial? A multicenter, prospective randomized controlled trial. J Hepatobiliary Pancreat Sci. 2015 Jul;22(7):551-7. doi: 10.1002/jhbp.244. Epub 2015 Apr 16. PMID 25881915

RESULTS

PARTICIPANT FLOW:
Groups:
- Drain Insertion: Laparoscopic cholecystectomy with drain insertion is performed in this arm.
  Laparoscopic cholecystectomy with drain insertion: In the drain insertion group, investigators use the closed suction drain through a lateral 5-mm trocar and placed it in Morrison's pouch.
Period: Overall Study
Arm/Group | Drain Insertion | no Drain Insertion
Started | 98 | 100
Completed | 94 | 99
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drain Insertion | no Drain Insertion | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15.6) | 50 (15.9) | 54 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 54 | 52 | 106
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 98 | 100 | 198

OUTCOME MEASURES:

1. Primary Outcome: Complication
Description: complication is subhepatic fluid collection with abscess or subhepatic hematoma or bile leakage.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | no Drain Insertion | Drain Insertion
Number analyzed (Participants) | 99 | 94
participants | 7 | 7

2. Secondary Outcome: Operative Time
Time Frame: 1day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Drain Insertion | no Drain Insertion
Number analyzed (Participants) | 94 | 99
minutes | 47.8 (17.7) | 43.1 (17.1)

3. Secondary Outcome: Postoperative Hospital Stay
Time Frame: 2weeks
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Drain Insertion | no Drain Insertion
Number analyzed (Participants) | 94 | 99
day | 2.5 (1.4) | 2.3 (0.8)

4. Secondary Outcome: Postoperative Pain Score
Description: Postoperative pain was estimated using the visual analog scale (VAS) from 0 (no pain) to 10 (worst pain imaginable) at 6, 24, and 48 hours after the operation.
Time Frame: 6hr after operation - 24hr after operation - 48hr after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drain Insertion | no Drain Insertion
Number analyzed (Participants) | 94 | 99
units on a scale
  6hr after operation | 5.0 (2.2) | 5.2 (2.4)
  24hr after operation | 3.9 (1.4) | 3.3 (2.0)
  48hr after operation | 2.1 (1.5) | 1.5 (1.4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Drain Insertion | no Drain Insertion
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/100
Other Adverse Events (participants affected / at risk) | 9/94 | 9/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drain Insertion (N=94) | no Drain Insertion (N=99)
wound infection (Skin and subcutaneous tissue disorders) | 4 | 3
voiding difficulty (Renal and urinary disorders) | 1 | 3
prolonged postoperative shoulder pain (General disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes